CLINICAL TRIAL: NCT04933513
Title: Development and Validation of a French Scale Measuring Preoperative Expectations of Parkinson's Disease Patients Candidate to Deep Brain Stimulation : the DBS-PS (Deep Brain Stimulation Perception Scale)
Brief Title: Development and Validation of a Scale Measuring Preoperative Expectations in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Bordeaux (Other); Poitiers University Hospital (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Mme Mylène MEYER, psychologist, PhD, Central Hospital, Nancy, France
Other Study IDs: 2020PI179
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease
Keywords: deep brain stimulation; preoperative expectations; DBS-PS; validation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative Parkinson' disease: pre DBS parkinson's disease patients responding to the DBS-PS scale preoperatively
  Interventions: Behavioral: pre DBS patients responding to the DBS-PS scale

INTERVENTIONS:
Behavioral: pre DBS patients responding to the DBS-PS scale — we propose to parkinson's disease patients selected for subthalamic deep brain stimulation to complete the DBS-PS scale preoperatively

SUMMARY:
Subthalamic nucleus deep brain stimulation (STN-DBS) has become a choice treatment for fluctuating Parkinson's disease (PD) patients, inducing remarkable improvement in motor symptoms. However, as PD is a complex neuropsychiatric disease, it has been hypothesized that in some patients, non-motor features, i.e. dysfunctional expectations for the result of neurosurgery, could interfere with postoperative result of DBS, even in case of motor improvement. Recent literature highlights the necessity to take these preoperative expectations into account, but to our knowledge, no specific scale investigating these cognitions in this PD-specific condition is available. So, the investigators developped the DBS-PS, a self-scale constructed to measure preoperative expectations for DBS, with 11 questions and visuo-analogical responses (1 to 10), theorically divided in three domains investigating the expectations concerning symptoms of PD, postoperative social-life and leisures, and postoperative familial and marital sphere. The investigators would like to validate this new-developped scale in the preoperative subthalamic nucleus deep brain stimulation population through patients recruited in the Predistim study, whereas the investigators did not recruite sufficiently patients through the PsyParkinson study, the one in which the DBS-PS scale was developed. The DBS-PS constitutes an interesting basis for the consideration of these cognitive and affective factors in preoperative PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients included in the Predistim study and having completed the DBS-PS scale during the preoperative phase

Exclusion Criteria:

* Parkinson's disease patients not included in the Predistim study or not having completed the DBS-PS scale during the preoperative phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Parkinson's disease patients selected for STN DBS and participating to the Predistim study
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Validation of the Deep-brain stimulation - perception scale (DBS-PS scale) | during the inclusion/baseline period of Predistim study
  Deep Brain Stimulation-Perception Scale completed by Parkinson's disease patients enrolled in the Predistim study; minimum scale score 0 - maximum scale score 50, for each sub-scores (3 dimensions) ; a higher score corresponding to higher expectations in the dimension, and a lower score coresponding to lower expectations in the dimension

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer M, Spitz E, Colnat-Coulbois S, Benatru I, Guehl D, Hainque E, Rolland AS, Corvol JC, Devilliers H, Schwan R, Devos D; PREDISTIM group. Development and validation of the DBS-PS (Deep Brain Stimulation-Perception Scale): Assessing parkinsonian patients' expectations to prevent post-operative disappointment? J Neurol Sci. 2024 Jul 15;462:123093. doi: 10.1016/j.jns.2024.123093. Epub 2024 Jun 13. PMID 38908172